CLINICAL TRIAL: NCT04971200
Title: Pilot Study Assessing the Effect of Tildrakizumab in Vitiligo
Acronym: TILDVIT-1227
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Premier Specialists, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-04-373
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Skin and Connective Tissue Diseases; Skin Diseases; Pigmentation Disorder; Hypopigmentation; Biologic; Vitiligo
Keywords: Tildrakizumab; non-segmental vitiligo; interleukin-23; IL-23; biological treatment; pilot study; Anti-Inflammatory Agents; Anti-Inflammatory Agents, Non-Steroidal; Vitiligo
MeSH Terms: conditions — Skin and Connective Tissue Diseases; Skin Diseases; Pigmentation Disorders; Hypopigmentation; Vitiligo | interventions — tildrakizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitiligo Patients on Tildrakizumab (Experimental)
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — 2 100mg subcutaneous injections Q4W

SUMMARY:
Vitiligo is a common acquired depigmentation disorder affecting approximately 2% of the world population. The purpose of this pilot study is to evaluate the effect and the safety of Tildrakizumab in adult participants with vitiligo.

DETAILED DESCRIPTION:
Tildrakizumab is a monoclonal antibody against interleukin (IL) 23, specifically anti-IL23p19. It is approved in the USA, Europe and Australia for psoriasis. The psoriasis dose is 100mg administered subcutaneously at weeks 0, 4 and every 12 weeks. Recent research has shown medications used to treat psoriasis may be effective in other immune mediated or autoimmune diseases such as vitiligo. With studies underway assessing the effect of Janus Kinase (JAK) inhibitors in psoriasis and vitiligo, this study seeks to determine if an IL-23 inhibitor is beneficial in halting disease progression and inducing repigmentation in vitiligo. There is some data to indicate that a higher dose of Tildrakizumab is effective for other autoimmune diseases such as psoriasis and hidradenitis suppurativa. For psoriasis, 200mg dosage was more effective than 100mg dosage. For hidradenitis suppurativa, a dosage of 200mg every 4 weeks was shown to be effective. Patients included in this study will start Tildrakizumab at a dosage of 200mg every 4 weeks for 6 months. There is a total of 8 visits involved in this study. Tildrakizumab is provided during visit 2, 3, 4, 5, 6, 7. Visit 1is a screening visit. At visit 1 and visit 8 no study drug will be provided.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of vitiligo
* Clinically stable vitiligo: defined as no new vitiligo patches and no enlargement of existing patches in previous 3 months.
* Able to provide voluntary, written, informed consent

Exclusion Criteria:

* Clinically active vitiligo: defined as new vitiligo patches or enlargement of existing patches in previous 3 months
* Concurrent skin disease in the study area
* Immunocompromise
* Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 12 weeks after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage repigmentation: Vitiligo Area Scoring Index (VASI) | Week 24
  Percentage repigmentation is assessed through change in score from baseline. Range 0-100. Higher score=greater depigmentation/worse
Percentage repigmentation: Vitiligo Extent Score (VES) | Week 24
  Percentage repigmentation is assessed through change in score from baseline. Range 0-100. Higher score=greater depigmentation/worse
Percentage repigmentation: Photographs | Week 24
  Percentage repigmentation is assessed through comparison of photographs of vitiligo lesions from baseline.

SECONDARY OUTCOMES:
Percentage repigmentation: Vitiligo Area Scoring Index (VASI) | Week 12
  Percentage repigmentation is assessed through change in score from baseline. Range 0-100. Higher score=greater depigmentation/worse
Percentage repigmentation: Vitiligo Extent Score (VES) | Week 12
  Percentage repigmentation is assessed through change in score from baseline. Range 0-100. Higher score=greater depigmentation/worse
Percentage repigmentation: Photographs | Week 12
  Percentage repigmentation is assessed through comparison of photographs of vitiligo lesions from baseline.
Time to repigmentation | through study treatment completion at 24-weeks
Change in Quality of Life score from baseline: Dermatology Life Quality Index (DLQI) | Baseline through week 12 and through study treatment completion at 24-weeks
  Used to assess treatment response on subject's quality of life. Range 0-30. Higher score=larger effect on patient's life/worse
Change in Quality of Life score from baseline: Patient Global Impression of Change (PGIC) | Baseline through week 12 and through study treatment completion at 24-weeks
  1-tem questionnaire designed to assess a subject's impression of disease improvement. 7 point Likert scale ranging from "Very much better" to "Very much worse" with "no change" in the middle. Range[1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderately better, 6-better/a definite improvement, 7-a great deal better]. Higher score=better impression of change/better
Change in Quality of Life score from baseline: Self-Assessment Vitiligo Extent Score (SA-VES) | Baseline through week 12 and through study treatment completion at 24-weeks
  Validated patient reported outcome measurement to provide information about disease extent and repigmentation. Range 0-100. Higher score=greater depigmentation/worse.
Adverse events | through study treatment completion at 24-weeks
  incidence and nature of any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dedee Murrell, MD, Principal Investigator — University of New South Wales
Locations (1):
- Premier Specialists Pty Ltd, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Jerjen R, Moodley A, Sinclair R. Repigmentation of acrofacial vitiligo with subcutaneous tildrakizumab. Australas J Dermatol. 2020 Nov;61(4):e446-e448. doi: 10.1111/ajd.13346. Epub 2020 May 21. No abstract available. PMID 32441048
- [Background] Vaccaro M, Cannavo SP, Imbesi S, Cristani M, Barbuzza O, Tigano V, Gangemi S. Increased serum levels of interleukin-23 circulating in patients with non-segmental generalized vitiligo. Int J Dermatol. 2015 Jun;54(6):672-4. doi: 10.1111/ijd.12392. Epub 2014 Nov 27. PMID 25427848
- [Background] Hu Y, Qi X, Hu Y, Lu Y, Liu K, Han X, Mao Z, Wu Z, Zhou X. Effects of CO2 fractional laser therapy on peripheral blood cytokines in patients with vitiligo. Dermatol Ther. 2019 Jul;32(4):e12992. doi: 10.1111/dth.12992. Epub 2019 Jun 17. PMID 31172649
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] van Geel N, Lommerts J, Bekkenk M, Wolkerstorfer A, Prinsen CAC, Eleftheriadou V, Taieb A, Picardo M, Ezzedine K, Speeckaert R. Development and Validation of the Vitiligo Extent Score (VES): an International Collaborative Initiative. J Invest Dermatol. 2016 May;136(5):978-984. doi: 10.1016/j.jid.2015.12.040. Epub 2016 Jan 28. PMID 26827762
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] van Geel N, Lommerts JE, Bekkenk MW, Prinsen CA, Eleftheriadou V, Taieb A, Picardo M, Ezzedine K, Wolkerstorfer A, Speeckaert R; international Vitiligo Score Working Group. Development and validation of a patient-reported outcome measure in vitiligo: The Self Assessment Vitiligo Extent Score (SA-VES). J Am Acad Dermatol. 2017 Mar;76(3):464-471. doi: 10.1016/j.jaad.2016.09.034. Epub 2016 Nov 22. PMID 27887798
- See also: Premier Specialists Dermatology — http://dermatologytrialsaustralia.com.au/